CLINICAL TRIAL: NCT02995005
Title: Prevention of Mother-to-child Transmission of Hepatitis B Virus: a One Arm, Open Label Intervention Study to Estimate the Optimal Timing of Tenofovir (TDF) in Pregnancy
Brief Title: Tenofovir in Early Pregnancy to Prevent Mother-to-child Transmission of Hepatitis B Virus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Thrasher Research Fund (Other); Shoklo Malaria Research Unit (Other); Chiang Mai University (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JHSPH-TDF; NCT03167229 (obsolete NCT alias)
Record Dates: First submitted 2016-12-08; First posted 2016-12-16 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2022-10

CONDITIONS: Hepatitis B
Keywords: mother to child transmission; hepatitis B; tenofovir
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Intervention Model Description: Single group study.
Masking Description: No masking, just one interventional group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tenofovir Disoproxil Fumarate (Experimental): Women early in pregnancy (end of first or beginning second trimester) will be treated with TDF to determine the efficacy of this strategy to bring >=95% of women to undetectable HBV DNA levels at delivery.
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — 300 mg daily
  Other Names: Viread

SUMMARY:
Mother-to-child transmission (MTCT) of hepatitis B virus (HBV) remains the major mode of transmission in most high and intermediate HBV endemic areas, despite existing WHO immunoprophylaxis recommendations. This immunoprophylaxis regimen, if given optimally, can prevent 75-80% of HBV MTCT, but optimal implementation is difficult because it requires administering monovalent HBV vaccine and hepatitis B immunoglobulin (HBIg) within 24 hours of birth. Due to the barriers of giving HBIg, the World Health Organization (WHO) states, "…owing to concerns related to supply, safety and cost, the use of HBIg is not feasible in most settings." Clearly, global control of HBV transmission will require improved MTCT prevention. Therefore, the investigators hypothesize that treating HBV early in pregnancy will lead to undetectable HBV DNA levels at delivery and prevention of MTCT of HBV without HBIg; a concept that has already been proven with HIV. Tenofovir disoproxil fumarate (TDF), an approved anti-HBV drug, is promising to prevent MTCT of HBV due to its high potency against hepatitis B and its safety record in pregnant women. A randomized, controlled clinical trial (RCT) will be necessary to determine if TDF given to HBV-infected pregnant women early in pregnancy plus vaccine to the newborn can decrease MTCT of HBV without HBIg. However, before embarking on a RCT, several critical knowledge gaps need to be addressed including the ideal timing for TDF initiation. The purpose of this proposal is to address these knowledge gaps.

DETAILED DESCRIPTION:
The investigators hypothesize that anti-HBV therapy given in the late first or early second trimester achieves undetectable HBV DNA at delivery in >=95% of pregnant women with chronic hepatitis B. The one-arm, open-label, interventional study aims: 1, To estimate the time to complete HBV DNA suppression (<100 IU/ml) in 170 HBV DNA positive women who start TDF in the late first or early second trimester; and to estimate the proportion of women with HBV DNA <100 IU/ml at delivery. 2, To address potential barriers to and the efficacy of implementing TDF in early pregnancy to prevent mother-to-child transmission of hepatitis B. The investigators will measure potential barriers to acceptability and effectiveness of this intervention: adherence, potential hepatitis B flares in mothers (safety), and the proportion of hepatitis B infections in the offspring at 1 year of age (efficacy).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 and over
* HBsAg positive
* In the 12th-20th week of pregnancy
* Willing to take TDF daily during pregnancy
* Providing written informed consent
* Plans to deliver at Shoklo Malaria Research Unit (SMRU)
* Able and willing to comply with study requirements

Exclusion Criteria:

* Anti-HIV positive
* Negative qualitative HBV DNA if HBeAg negative
* On immunosuppressive therapy
* Elevated creatinine
* History of kidney disease
* Short cervix
* History of pregnancy complications or prior pre-term labor

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
The time (from inclusion through delivery; up to 6 months) to HBV DNA suppression (<100 IU/ml) | Up to 9 months
  HBV DNA will be monitored every month
The proportion of women with undetectable HBV DNA at delivery | At delivery
  HBV DNA will be monitored at delivery.

SECONDARY OUTCOMES:
Proportion of hepatitis B flares in mothers postpartum | Monthly measured for 3 months after stopping TDF.
  All women will continue on study for 3 months after stopping TDF to measure their alanine aminotransferase (ALT) and aspartate aminotransferase (AST) monthly to detect a flare, which will be defined as >5x baseline or >10x the upper limit of normal. If at the end of the 3 months, there has been no change in ALT and AST, then the mothers will be discharged from the study. If there is an increase in liver enzymes but not a true flare, they will be followed for an additional 3 months with monthly ALT testing.
The proportion of women who adhered to TDF treatment during the course of the study (from inclusion through 1 month after delivery; up to 7 months; drug levels) | Up to 9 months
  Measurement of tenofovir drug levels
The proportion of women who adhered to TDF treatment during the course of the study (from inclusion through 1 month after delivery; up to 7 months; drug accountability) | Up to 9 months
  Drug accountability using standard methods (subtracting the number of tablets left from the number of tablets distributed).
The proportion of women who adhered to TDF treatment during the course of the study (from inclusion through 1 month after delivery; up to 7 months; questionnaire) | Up to 9 months
  All women will be surveyed at monthly visits and at birth to measure adherence including actionable barriers.
The proportion of hepatitis B infections in the offspring at 1 year of age | Between month 2 and 12 month
  Testing for HBsAg in children between 2 and 12 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Ehrhardt, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The investigators are currently developing an individual participant data (IPD) sharing plan.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available 6 months after publication of the main report.
Access Criteria: Permission by corresponding author

REFERENCES:
- [Background] Lee WM. Hepatitis B virus infection. N Engl J Med. 1997 Dec 11;337(24):1733-45. doi: 10.1056/NEJM199712113372406. No abstract available. PMID 9392700
- [Background] Lavanchy D. Worldwide epidemiology of HBV infection, disease burden, and vaccine prevention. J Clin Virol. 2005 Dec;34 Suppl 1:S1-3. doi: 10.1016/s1386-6532(05)00384-7. PMID 16461208
- [Background] Ranger-Rogez S, Denis F. Hepatitis B mother--to--child transmission. Expert Rev Anti Infect Ther. 2004 Feb;2(1):133-45. doi: 10.1586/14787210.2.1.133. PMID 15482178
- [Background] Chang MH. Natural history of hepatitis B virus infection in children. J Gastroenterol Hepatol. 2000 May;15 Suppl:E16-9. doi: 10.1046/j.1440-1746.2000.02096.x. PMID 10921376
- [Background] Wen WH, Chang MH, Zhao LL, Ni YH, Hsu HY, Wu JF, Chen PJ, Chen DS, Chen HL. Mother-to-infant transmission of hepatitis B virus infection: significance of maternal viral load and strategies for intervention. J Hepatol. 2013 Jul;59(1):24-30. doi: 10.1016/j.jhep.2013.02.015. Epub 2013 Feb 26. PMID 23485519
- [Background] Chien YC, Jan CF, Kuo HS, Chen CJ. Nationwide hepatitis B vaccination program in Taiwan: effectiveness in the 20 years after it was launched. Epidemiol Rev. 2006;28:126-35. doi: 10.1093/epirev/mxj010. Epub 2006 Jun 16. PMID 16782778
- [Background] Xu H, Zeng T, Liu JY, Lei Y, Zhong S, Sheng YJ, Zhou Z, Ren H. Measures to reduce mother-to-child transmission of Hepatitis B virus in China: a meta-analysis. Dig Dis Sci. 2014 Feb;59(2):242-58. doi: 10.1007/s10620-013-2918-0. Epub 2013 Nov 6. PMID 24193353
- [Background] Xu DZ, Yan YP, Choi BC, Xu JQ, Men K, Zhang JX, Liu ZH, Wang FS. Risk factors and mechanism of transplacental transmission of hepatitis B virus: a case-control study. J Med Virol. 2002 May;67(1):20-6. doi: 10.1002/jmv.2187. PMID 11920813
- [Background] Shao ZJ, Zhang L, Xu JQ, Xu DZ, Men K, Zhang JX, Cui HC, Yan YP. Mother-to-infant transmission of hepatitis B virus: a Chinese experience. J Med Virol. 2011 May;83(5):791-5. doi: 10.1002/jmv.22043. Epub 2011 Feb 25. PMID 21360547
- [Background] Chen DS. Hepatitis B vaccination: The key towards elimination and eradication of hepatitis B. J Hepatol. 2009 Apr;50(4):805-16. doi: 10.1016/j.jhep.2009.01.002. Epub 2009 Feb 3. PMID 19231008
- [Background] Wiseman E, Fraser MA, Holden S, Glass A, Kidson BL, Heron LG, Maley MW, Ayres A, Locarnini SA, Levy MT. Perinatal transmission of hepatitis B virus: an Australian experience. Med J Aust. 2009 May 4;190(9):489-92. doi: 10.5694/j.1326-5377.2009.tb02524.x. PMID 19413519
- [Background] Tran TT. Management of hepatitis B in pregnancy: weighing the options. Cleve Clin J Med. 2009 May;76 Suppl 3:S25-9. doi: 10.3949/ccjm.76.s3.06. PMID 19465706
- [Background] del Canho R, Grosheide PM, Mazel JA, Heijtink RA, Hop WC, Gerards LJ, de Gast GC, Fetter WP, Zwijneberg J, Schalm SW. Ten-year neonatal hepatitis B vaccination program, The Netherlands, 1982-1992: protective efficacy and long-term immunogenicity. Vaccine. 1997 Oct;15(15):1624-30. doi: 10.1016/s0264-410x(97)00080-7. PMID 9364693
- [Background] Read JS. Prevention of mother-to-child transmission of HIV: antiretroviral strategies. Clin Perinatol. 2010 Dec;37(4):765-76, viii. doi: 10.1016/j.clp.2010.08.007. PMID 21078449
- [Background] Warszawski J, Tubiana R, Le Chenadec J, Blanche S, Teglas JP, Dollfus C, Faye A, Burgard M, Rouzioux C, Mandelbrot L; ANRS French Perinatal Cohort. Mother-to-child HIV transmission despite antiretroviral therapy in the ANRS French Perinatal Cohort. AIDS. 2008 Jan 11;22(2):289-99. doi: 10.1097/QAD.0b013e3282f3d63c. PMID 18097232
- [Background] Garcia PM, Kalish LA, Pitt J, Minkoff H, Quinn TC, Burchett SK, Kornegay J, Jackson B, Moye J, Hanson C, Zorrilla C, Lew JF. Maternal levels of plasma human immunodeficiency virus type 1 RNA and the risk of perinatal transmission. Women and Infants Transmission Study Group. N Engl J Med. 1999 Aug 5;341(6):394-402. doi: 10.1056/NEJM199908053410602. PMID 10432324
- [Background] Burk RD, Hwang LY, Ho GY, Shafritz DA, Beasley RP. Outcome of perinatal hepatitis B virus exposure is dependent on maternal virus load. J Infect Dis. 1994 Dec;170(6):1418-23. doi: 10.1093/infdis/170.6.1418. PMID 7995980
- [Background] Lai CL, Gane E, Liaw YF, Hsu CW, Thongsawat S, Wang Y, Chen Y, Heathcote EJ, Rasenack J, Bzowej N, Naoumov NV, Di Bisceglie AM, Zeuzem S, Moon YM, Goodman Z, Chao G, Constance BF, Brown NA; Globe Study Group. Telbivudine versus lamivudine in patients with chronic hepatitis B. N Engl J Med. 2007 Dec 20;357(25):2576-88. doi: 10.1056/NEJMoa066422. PMID 18094378
- [Background] Gordon SC, Krastev Z, Horban A, Petersen J, Sperl J, Dinh P, Martins EB, Yee LJ, Flaherty JF, Kitrinos KM, Rustgi VK, Marcellin P. Efficacy of tenofovir disoproxil fumarate at 240 weeks in patients with chronic hepatitis B with high baseline viral load. Hepatology. 2013 Aug;58(2):505-13. doi: 10.1002/hep.26277. Epub 2013 May 3. PMID 23364953
- [Background] Pan CQ, Mi LJ, Bunchorntavakul C, Karsdon J, Huang WM, Singhvi G, Ghany MG, Reddy KR. Tenofovir disoproxil fumarate for prevention of vertical transmission of hepatitis B virus infection by highly viremic pregnant women: a case series. Dig Dis Sci. 2012 Sep;57(9):2423-9. doi: 10.1007/s10620-012-2187-3. Epub 2012 Apr 29. PMID 22543886
- [Background] European Association For The Study Of The Liver. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012 Jul;57(1):167-85. doi: 10.1016/j.jhep.2012.02.010. Epub 2012 Mar 20. No abstract available. PMID 22436845
- [Background] Pan CQ, Duan ZP, Bhamidimarri KR, Zou HB, Liang XF, Li J, Tong MJ. An algorithm for risk assessment and intervention of mother to child transmission of hepatitis B virus. Clin Gastroenterol Hepatol. 2012 May;10(5):452-9. doi: 10.1016/j.cgh.2011.10.041. Epub 2011 Nov 9. PMID 22079509
- [Background] Li XM, Yang YB, Hou HY, Shi ZJ, Shen HM, Teng BQ, Li AM, Shi MF, Zou L. Interruption of HBV intrauterine transmission: a clinical study. World J Gastroenterol. 2003 Jul;9(7):1501-3. doi: 10.3748/wjg.v9.i7.1501. PMID 12854150
- [Background] Buti M, Tsai N, Petersen J, Flisiak R, Gurel S, Krastev Z, Aguilar Schall R, Flaherty JF, Martins EB, Charuworn P, Kitrinos KM, Subramanian GM, Gane E, Marcellin P. Seven-year efficacy and safety of treatment with tenofovir disoproxil fumarate for chronic hepatitis B virus infection. Dig Dis Sci. 2015 May;60(5):1457-64. doi: 10.1007/s10620-014-3486-7. Epub 2014 Dec 23. PMID 25532501
- [Background] Lim YS, Byun KS, Yoo BC, Kwon SY, Kim YJ, An J, Lee HC, Lee YS. Tenofovir monotherapy versus tenofovir and entecavir combination therapy in patients with entecavir-resistant chronic hepatitis B with multiple drug failure: results of a randomised trial. Gut. 2016 May;65(5):852-60. doi: 10.1136/gutjnl-2014-308353. Epub 2015 Jan 16. PMID 25596179
- [Background] Han GR, Jiang HX, Yue X, Ding Y, Wang CM, Wang GJ, Yang YF. Efficacy and safety of telbivudine treatment: an open-label, prospective study in pregnant women for the prevention of perinatal transmission of hepatitis B virus infection. J Viral Hepat. 2015 Sep;22(9):754-62. doi: 10.1111/jvh.12379. Epub 2015 Jan 12. PMID 25641421
- [Background] Zhang H, Pan CQ, Pang Q, Tian R, Yan M, Liu X. Telbivudine or lamivudine use in late pregnancy safely reduces perinatal transmission of hepatitis B virus in real-life practice. Hepatology. 2014 Jan 27. doi: 10.1002/hep.27034. Online ahead of print. PMID 25227594
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B: update 2009. Hepatology. 2009 Sep;50(3):661-2. doi: 10.1002/hep.23190. No abstract available. PMID 19714720
- [Background] Liu Y, Wang M, Yao S, Yuan J, Lu J, Li H, Zeng W, Deng Y, Zou R, Li J, Xiao J. Efficacy and safety of telbivudine in different trimesters of pregnancy with high viremia for interrupting perinatal transmission of hepatitis B virus. Hepatol Res. 2016 Mar;46(3):E181-8. doi: 10.1111/hepr.12525. Epub 2015 May 21. PMID 25869545
- [Background] Van Damme L, Corneli A, Ahmed K, Agot K, Lombaard J, Kapiga S, Malahleha M, Owino F, Manongi R, Onyango J, Temu L, Monedi MC, Mak'Oketch P, Makanda M, Reblin I, Makatu SE, Saylor L, Kiernan H, Kirkendale S, Wong C, Grant R, Kashuba A, Nanda K, Mandala J, Fransen K, Deese J, Crucitti T, Mastro TD, Taylor D; FEM-PrEP Study Group. Preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2012 Aug 2;367(5):411-22. doi: 10.1056/NEJMoa1202614. Epub 2012 Jul 11. PMID 22784040
- [Background] Marrazzo JM, Ramjee G, Richardson BA, Gomez K, Mgodi N, Nair G, Palanee T, Nakabiito C, van der Straten A, Noguchi L, Hendrix CW, Dai JY, Ganesh S, Mkhize B, Taljaard M, Parikh UM, Piper J, Masse B, Grossman C, Rooney J, Schwartz JL, Watts H, Marzinke MA, Hillier SL, McGowan IM, Chirenje ZM; VOICE Study Team. Tenofovir-based preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2015 Feb 5;372(6):509-18. doi: 10.1056/NEJMoa1402269. PMID 25651245
- [Background] Siberry GK, Jacobson DL, Kalkwarf HJ, Wu JW, DiMeglio LA, Yogev R, Knapp KM, Wheeler JJ, Butler L, Hazra R, Miller TL, Seage GR 3rd, Van Dyke RB, Barr E, Davtyan M, Mofenson LM, Rich KC; Pediatric HIV/AIDS Cohort Study. Lower Newborn Bone Mineral Content Associated With Maternal Use of Tenofovir Disoproxil Fumarate During Pregnancy. Clin Infect Dis. 2015 Sep 15;61(6):996-1003. doi: 10.1093/cid/civ437. Epub 2015 Jun 9. PMID 26060285
- [Background] Nguyen V, Tan PK, Greenup AJ, Glass A, Davison S, Samarasinghe D, Holdaway S, Strasser SI, Chatterjee U, Jackson K, Locarnini SA, Levy MT. Anti-viral therapy for prevention of perinatal HBV transmission: extending therapy beyond birth does not protect against post-partum flare. Aliment Pharmacol Ther. 2014 May;39(10):1225-34. doi: 10.1111/apt.12726. Epub 2014 Mar 25. PMID 24666381
- [Background] Mondou E, Sorbel J, Anderson J, Mommeja-Marin H, Rigney A, Rousseau F. Posttreatment exacerbation of hepatitis B virus (HBV) infection in long-term HBV trials of emtricitabine. Clin Infect Dis. 2005 Sep 1;41(5):e45-7. doi: 10.1086/432581. Epub 2005 Jul 20. PMID 16080074
- [Background] Thio CL, Guo N, Xie C, Nelson KE, Ehrhardt S. Global elimination of mother-to-child transmission of hepatitis B: revisiting the current strategy. Lancet Infect Dis. 2015 Aug;15(8):981-5. doi: 10.1016/S1473-3099(15)00158-9. Epub 2015 Jul 2. PMID 26145195
- [Background] Ehrhardt S, Xie C, Guo N, Nelson K, Thio CL. Breastfeeding while taking lamivudine or tenofovir disoproxil fumarate: a review of the evidence. Clin Infect Dis. 2015 Jan 15;60(2):275-8. doi: 10.1093/cid/ciu798. Epub 2014 Oct 13. PMID 25313254
- [Background] Hahn SR, Park J, Skinner EP, Yu-Isenberg KS, Weaver MB, Crawford B, Flowers PW. Development of the ASK-20 adherence barrier survey. Curr Med Res Opin. 2008 Jul;24(7):2127-38. doi: 10.1185/03007990802174769. Epub 2008 Jun 12. PMID 18554431
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Beigi R, Noguchi L, Parsons T, Macio I, Kunjara Na Ayudhya RP, Chen J, Hendrix CW, Masse B, Valentine M, Piper J, Watts DH. Pharmacokinetics and placental transfer of single-dose tenofovir 1% vaginal gel in term pregnancy. J Infect Dis. 2011 Nov 15;204(10):1527-31. doi: 10.1093/infdis/jir562. Epub 2011 Sep 19. PMID 21930612
- [Background] Hendrix CW, Chen BA, Guddera V, Hoesley C, Justman J, Nakabiito C, Salata R, Soto-Torres L, Patterson K, Minnis AM, Gandham S, Gomez K, Richardson BA, Bumpus NN. MTN-001: randomized pharmacokinetic cross-over study comparing tenofovir vaginal gel and oral tablets in vaginal tissue and other compartments. PLoS One. 2013;8(1):e55013. doi: 10.1371/journal.pone.0055013. Epub 2013 Jan 30. PMID 23383037
- [Background] Choopanya K, Martin M, Suntharasamai P, Sangkum U, Mock PA, Leethochawalit M, Chiamwongpaet S, Kitisin P, Natrujirote P, Kittimunkong S, Chuachoowong R, Gvetadze RJ, McNicholl JM, Paxton LA, Curlin ME, Hendrix CW, Vanichseni S; Bangkok Tenofovir Study Group. Antiretroviral prophylaxis for HIV infection in injecting drug users in Bangkok, Thailand (the Bangkok Tenofovir Study): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2013 Jun 15;381(9883):2083-90. doi: 10.1016/S0140-6736(13)61127-7. Epub 2013 Jun 13. PMID 23769234
- [Background] Seserko LA, Emory JF, Hendrix CW, Marzinke MA. The development and validation of an UHPLC-MS/MS method for the rapid quantification of the antiretroviral agent dapivirine in human plasma. Bioanalysis. 2013 Nov;5(22):2771-83. doi: 10.4155/bio.13.256. PMID 24256358
- [Background] Minnis AM, Gandham S, Richardson BA, Guddera V, Chen BA, Salata R, Nakabiito C, Hoesley C, Justman J, Soto-Torres L, Patterson K, Gomez K, Hendrix CW. Adherence and acceptability in MTN 001: a randomized cross-over trial of daily oral and topical tenofovir for HIV prevention in women. AIDS Behav. 2013 Feb;17(2):737-47. doi: 10.1007/s10461-012-0333-8. PMID 23065145
- [Background] Anderson PL, Glidden DV, Liu A, Buchbinder S, Lama JR, Guanira JV, McMahan V, Bushman LR, Casapia M, Montoya-Herrera O, Veloso VG, Mayer KH, Chariyalertsak S, Schechter M, Bekker LG, Kallas EG, Grant RM; iPrEx Study Team. Emtricitabine-tenofovir concentrations and pre-exposure prophylaxis efficacy in men who have sex with men. Sci Transl Med. 2012 Sep 12;4(151):151ra125. doi: 10.1126/scitranslmed.3004006. PMID 22972843
- [Background] Zhao Z, Ding M, Hu Z, Dai Q, Satija A, Zhou A, Xu Y, Zhang X, Hu FB, Xu H. Trajectories of length, weight, and bone mineral density among preterm infants during the first 12 months of corrected age in China. BMC Pediatr. 2015 Aug 5;15:91. doi: 10.1186/s12887-015-0396-6. PMID 26242232
- [Derived] Bierhoff M, Nelson KE, Guo N, Jia Y, Angkurawaranon C, Jittamala P, Carrara V, Watthanaworawit W, Ling C, Tongprasert F, van Vugt M, Rijken M, Nosten F, McGready R, Ehrhardt S, Thio CL. Prevention of mother-to-child transmission of hepatitis B virus: protocol for a one-arm, open-label intervention study to estimate the optimal timing of tenofovir in pregnancy. BMJ Open. 2020 Sep 13;10(9):e038123. doi: 10.1136/bmjopen-2020-038123. PMID 32928858
- [Derived] Bierhoff M, Rijken MJ, Yotyingaphiram W, Pimanpanarak M, van Vugt M, Angkurawaranon C, Nosten F, Ehrhardt S, Thio CL, McGready R. Tenofovir for prevention of mother to child transmission of hepatitis B in migrant women in a resource-limited setting on the Thailand-Myanmar border: a commentary on challenges of implementation. Int J Equity Health. 2020 Sep 10;19(1):156. doi: 10.1186/s12939-020-01268-3. PMID 32912268